CLINICAL TRIAL: NCT05495776
Title: Prospective Multicenter Registry Study to Assess the Frequency of Lynch Syndrome Among Patients With Colorectal Cancer
Acronym: MSIRus22
Status: Recruiting | Type: Observational
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Collaborators: The Loginov MCSC MHD (Unknown); Pirogov National Medical and Surgical Center (Unknown); Moscow City Oncological Hospital No. 62 MHD (Unknown); City Clinical Oncological Hospital No. 1 MHD (Unknown); MMCC Kommunarka MHD (Unknown); D.D. Pletnev City Clinical Hospital MHD (Unknown); Botkin Hospital MHD (Unknown); Clinic K+31 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01082022
Record Dates: First submitted 2022-07-29; First posted 2022-08-10 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Lynch Syndrome; Hereditary Colorectal Cancer; MSI
Keywords: Colorectal Cancer; Lynch Syndrome; Hereditary Colorectal Cancer; MSI; Frequency
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — In case of microsatellite instability/deficiency in the repair system of unpaired bases, venous blood will be taken 4 ml into a test tube with EDTA with freezing at -20 * C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colorectal cancer: Patients with colon adenocarcinoma who have not previously received antitumor treatment (chemo/radiation therapy) for a currently detected tumor

SUMMARY:
Prospective multicenter registry study to assess the frequency of Lynch syndrome among patients with colorectal cancer in Russia

DETAILED DESCRIPTION:
Blood and tumor samples will be obtained from enrolled patients. 4 ml of venous blood samples will be taken into a tube with EDTA and stored at -20 0C. Tumor samples will be taken during endoscopy or surgical treatment, embedded in paraffin and stored at room temperature.

Microsatellite instability in the tumor tissue will be determined by any method available in the participating center (immunohistochemical or molecular genetic study). In case of detection of microsatellite instability/deficiency in the repair system of unpaired bases blood samples will be analyzed for the fact that germinal mutations in the DNA mismatch repair genes.

Patients will be followed up for 5 years after enrollment. During follow up correlation of spectrum of germinal mutations with clinical data, effectiveness of therapy with immune checkpoint inhibitors, the spectrum of malignant neoplasms in the families of patients with Lynch syndrome, the impact of the presence of microsatellite instability/deficiency in the DNA mismatch repair genes on treatment tactics in the Russian Federation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent;
* Patients with histologically verified colon adenocarcinoma or patients with histologically verified synchronous neoplasms who have not previously received treatment for a second tumor;
* Age ≥ 18 years;
* Absence of antitumor treatment for a real tumor (it is allowed to include patients who have a history of antitumor treatment for other malignant tumors, if the period after treatment is more than 12 months).
* The ability of the patient, according to the Researcher, to fulfill the requirements of the Protocol;

Exclusion Criteria:

- Patients receiving chemotherapy or radiotherapy for colon cancer at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon adenocarcinoma who have not previously received antitumor treatment (chemo/radiation therapy) for a currently detected tumor
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of microsatellite instability and Lynch syndrome | up to 5 years
  To assess the frequency of microsatellite instability and Lynch syndrome in the population of patients with colorectal cancer in the Russian Federation.

SECONDARY OUTCOMES:
Frequency of occurrence of microsatellite instability/deficiency | up to 5 years
  Assessment of the frequency of occurrence of microsatellite instability/deficiency in the repair system of unpaired bases in second tumors in patients with colorectal cancer of various stages.
Spectrum of germinal mutations in Lynch syndrome | up to 5 years
  The mlh1, msh2, msh6, pms2 and epcam genes will be examined for the presence of all types of pathogenic variants in patients with MSI in colon tumor. The possible correlation of gene-phenotype and pathogenic variants of each gene-phenotype will also be studied. To detect MSI in a tumor sample, need to do the fragment analysis (markers NR21, NR24, NR27, BAT25, BAT26). Рatients with MSI in the tumor will have DNA diagnostics of MMR EPCAM genes by sequencing and MLPA . The MMR and EPCAM genes will be examined in DNA isolated from blood lymphocytes.
Spectrum of malignant neoplasms | up to 5 years
  The family history of all oncological diseases will be studied to find out the main target organs of patients with Lynch syndrome in Russia
Effectiveness of therapy with immune checkpoint inhibitors | up to 5 years
  The frequency will be compared: the frequency of objective response rate (RECIST 1.1) while using immune checkpoint inhibitors in metastatic colon cancer and microsatellite instability associated/not associated with Lynch syndrome
Impact of the presence of microsatellite instability/deficiency | up to 5 years
  The frequency of adjuvant chemotherapy in stages II-III of colon cancer in the presence of microsatellite instability / deficiency in the repair system of unpaired bases in real clinical practice will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Tsukanov, PhD, Principal Investigator — Head of the Department of Laboratory Genetics
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Before the start of the study, at the initiating visit, the monitor, together with the researchers and their staff, will review the protocol and the CRF. During the study, the monitor will regularly communicate remotely with the research center and check the process of inclusion of patients, the completeness of maintaining medical records of patients, the correctness of filling out the CRF. The researcher must provide the monitor with access to the relevant hospital documentation and other medical records to verify their compliance with the data recorded in the IRC. The data identifying the patient's identity will remain confidential.
Supporting Information: CSR
Time Frame: 6 months after completion of the study
Access Criteria: upon the request